CLINICAL TRIAL: NCT06658483
Title: Investigation of the Turkish Validity and Reliability of the Hand ScleroDerma Lived Experience Scale (HAnDE Scale) Questionnaire in Individuals with Systemic Sclerosis
Brief Title: Hand ScleroDerma Lived Experience Scale in Individuals with Systemic Sclerosis
Status: Enrolling by invitation | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Zülal TATAR, researcher, Pamukkale University
Other Study IDs: Validity and Reliability
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Systemic Sclerosis (SSc); Hand Function
MeSH Terms: conditions — Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study was to examine the Turkish validity and reliability of the Hand scleroDerma lived Experience Scale (HAnDE Scale) Questionnaire in individuals with SSc.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Systemic Sclerosis by a rheumatologist
* Being 18 years of age or older,

Exclusion Criteria:

* Presence of neurological disease
* Presence of any orthopedic problem that will affect functionality
* Presence of orthopedic surgery history
* Inability to speak or understand Turkish fluently.
* Presence of psychiatric disease that will affect cooperation.
* Severe neurological disease that will affect hand functions (peripheral nerve lesion, trauma, operation, cerebrovascular accident).
* Heart failure and lung pathology that will affect daily living activities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include individuals aged 18 and older who are receiving treatment for Systemic Sclerosis at two university hospital in Turkey, and meet the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-07-24 (Estimated); Study Completion 2025-07-24 (Estimated)

PRIMARY OUTCOMES:
Hand ScleroDerma Lived Experience Scale (HAnDE Scale) Questionnaire | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  The scale consists of 18 items regarding the patient-reported status of hand function in individuals with SSc. Each response ranges from 0 to 4. 0 means 'completely disagree' and 4 means 'completely agree'. The higher the scale score, the worse the experience with the hand

SECONDARY OUTCOMES:
Hand Mobility in Scleroderma Test | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  It is a functional test that evaluates hand mobility. It evaluates 4 specific movements for the hand. These are extension, flexion, finger abduction and wrist dorsal extension. Various objects are used for evaluations, including cutting tool handles, pens, coffee packages, coils of rope, milk packages and tables. Each movement is scored between 0 and 3. 0 is used for being able to perform the movement normally and 3 for being completely unable to perform it. The total score is calculated by adding the scores for each movement and the highest score is 12.
Scleroderma Skin Involvement: Patient-Reported Outcomes | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Scleroderma Skin Involvement: Patient-Reported Outcomes was developed to assess skin-related quality of life in patients with systemic sclerosis. SSPRO consists of four domains: physical impact, emotional impact, physical limitation, and social impact, and consists of 18 items in total. Items are rated on a 6-point scale from no disability (0 points) to severe disability (6 points). The scores are added together to calculate a final score (0 to 108 points). A lower score indicates a much better quality of life
Modified Rodnan Skin Thickness Score | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  This method used to assess skin thickness in SSc. The Modified Rodnan Skin Thickness Score assesses skin thickness from 17 body regions. A score of 0 indicates normal skin thickness, 1 indicates mild skin thickness, 2 indicates moderate skin thickness, and 3 indicates severe skin thickness; a score of 3 indicates that the skin layers cannot be made between two fingers. The score is calculated by summing the scores from all 17 regions (range 0-51)
Scleroderma Health Assessment Questionnaire | Evaluations started immediately after receiving ethics committee approval and will be completed within 6 months, which is the study period.
  Used to assess disease activity. It has 20 items in 8 sections assessing physical disability. In addition, Raynaud phenomenon, digital ulcers, pulmonary and gastrointestinal symptoms are assessed according to the Visual Analog Scale, which is scored between "0" and "10". VAS is scored between 0 and 3 by multiplying by 0.2

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Inonu University, Malatya, Malatya
  - Pamukkale University, Denizli